CLINICAL TRIAL: NCT06388551
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, SAD Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Oral LPM526000133 Fumarate Capsules (LY03017) in Healthy Adult Subjects.
Brief Title: A Phase 1, SAD Study to Evaluate the Safety and Tolerability of LY03017
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03017/CT-CHN-101
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hallucinations and Delusions Associated With Alzheimer's Disease Psychosis; Hallucinations and Delusions Associated With Parkinson Disease Psychosis; Negative Symptoms of Schizophrenia
MeSH Terms: conditions — Hallucinations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY03017 (Experimental): Ascending single oral doses of LY03017 in healthy adult subjects
  Interventions: Drug: LY03017
- Placebo (Placebo Comparator): LY03017-Placebo
  Interventions: Drug: LY03017-Placebo

INTERVENTIONS:
Drug: LY03017 — single dose, administered orally
  Other Names: LPM526000133 Fumarate Capsules
  Arms: LY03017
Drug: LY03017-Placebo — single dose, administered orally
  Arms: Placebo

SUMMARY:
This is a phase 1，randomized, double-blind, placebo-controlled, SAD study to evaluate the safety, tolerability and pharmacokinetics of oral LPM526000133 Fumarate Capsules (LY03017) in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject who voluntarily participate and sign the informed consent form.
* Healthy male/female volunteers aged ≥18 and ≤ 45 years.
* Body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women, and body mass index (BMI) ≥18.5 and < 26.0 kg/m2.
* Able to comply with the lifestyle restrictions.

Exclusion Criteria:

* Subject has a history of allergy to any component of the investigational drug or similar drugs, or allergic constitution.
* Subject has a current or past medical history that may affect the clinical trial or dysfunction, including but not limited to the past or current respiratory system, circulatory system, digestive system, urinary system, reproductive system, nervous system, endocrine system, immune system, motor system, blood system, psychiatry/ psychology, dermatology and other clinically serious diseases or chronic diseases; or any other diseases that may interfere with the test results.
* Any surgical condition or condition may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects.
* Subject has a history of surgery within 3 months prior to administration, or failure to recover from surgery, or having an expected surgical plan during the trial.
* Subject has abnormal vital signs, laboratory abnormalities, and ECGs.
* Subject has used any of over-the-counter products within 7 days or prescription medications within 28 days prior to dosing.
* Subject positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), or syphilis seroreactivity (Trust).
* Subject has a history of alcohol abuse within 1 year or positive alcohol breath test results.
* Subject has a history of substance abuse within 1 year or a positive urine drug screen.
* Subject who has daily smoking of ≥ 5 cigarettes within 3 months.
* Subject who has special requirements for food, cannot comply with the unified diet or have dysphagia.
* Subject who has consumption of special diet (such as grapefruit, chocolate, coffee, xanthine-rich foods/drinks) within 48 hours prior to dosing and/or subject who has excessive daily consumption of tea, coffee, grapefruit juice, caffeinated beverages for nearly 3 months.
* Subject who has participated in other clinical trials within 3 months before administration.
* Subject has used blood products or being blood donor or blood loss within 3 months.
* Pregnant, lactating women, or positive pregnancy test.
* Subject who refusal to contraception, or plan to donate sperm or ovums.
* Subject who has a history of needle or blood faintness.
* Subject directly involved in this clinical trial.
* Poor compliance or other conditions which would make participation in the study unsuitable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | up to 216 hours

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of LPM526000133 in plasma | up to 216 hours
Time to maximum observed concentration (Tmax) of LPM526000133 in plasma | up to 216 hours
The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of LPM526000133 in plasma | up to 216 hours
Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC[0-last]) of LPM526000133 in plasma | up to 216 hours
Apparent terminal elimination half-life (t1/2) of LPM526000133 in plasma | up to 216 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China